CLINICAL TRIAL: NCT05796921
Title: Lacticaseibacillus Rhamnosus CA15 (DSM 33960) Strain as a New Driver in Restoring the Normal Vaginal Microbiota: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Lacticaseibacillus Rhamnosus CA15 (DSM 33960) Strain as a New Driver in Restoring the Normal Vaginal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agnese Maria Chiara Rapisarda (Other)
Collaborators: ProBioEtna (Unknown)
Responsible Party: Sponsor-Investigator, Agnese Maria Chiara Rapisarda, doctor, Universita degli Studi di Catania
Organization: Universita degli Studi di Catania (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 163/2022/PO
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Bacterial Vaginosis; Candidosis Vaginal; Urinary Tract Infections
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: randomized double-blind placebo-control
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): 1 daily capsule of the Lacticaseibacillus rhamnosus CA15 (DSM 33960) probiotic strain (10 billion of Colony Forming Units/capsule) for 10 days
  Interventions: Dietary Supplement: Lacticaseibacillus rhamnosus CA15 (DSM 33960) probiotic strain
- Placebo (Placebo Comparator): 1 daily capsule of placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lacticaseibacillus rhamnosus CA15 (DSM 33960) probiotic strain — Patients allocated to the probiotic arm will take the dietary supplement, containing 10 billion of the Lacticaseibacillus rhamnosus CA15 (DSM 33960) probiotic strain, once a day for 10 consecutive days.
  Other Names: probiotic CA15
  Arms: Active
Dietary Supplement: placebo — Patients allocated to placebo arm will take placebo capsules once a day for 10 consecutive days.
  Arms: Placebo

SUMMARY:
The aim of the present randomized double-blind placebo-controlled trial is to evaluate the efficacy of a probiotic formulation, containing the probiotic strain Lacticaseibacillus rhamnosus CA15 (DSM 33960), in the treatment of vaginal dysbiosis in terms of: (i) modulation of the microbiota (increase of lactobacilli and decrease of pathogens), (ii) reduction of clinical signs of inflammation, (iii) improvement of quality of life.

DETAILED DESCRIPTION:
The aim of the present randomized double-blind placebo-controlled study is to evaluate the ability of the potential probiotic Lacticaseibacillus rhamnosus CA15 (DSM 33960) strain, orally administrated, to balance the vaginal microbiota of women with vaginal dysbiosis. Two hundred women, with signs and symptoms of vaginal dysbiosis, are recruited and randomly allocated to receive oral capsules containing the L. rhamnosus CA15 (DSM 33960) strain or placebo once daily for 10 days. Clinical and microbiological parameters are evaluated in three scheduled appointments: at baseline (T0), 10 days after the start of the treatment (T1), and 30 days after the end of the treatment (T2). In addition, at baseline (T0) and 30 days after the end of the treatment (T2), the quality of life will be evaluated through a quality of life assessment questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one vaginal sign or symptom (leucorrhoea, burning, itching, subjective vaginal discomfort);
* Presence of at least 3 Amsel criteria;
* Nugent score greater than 7;
* Lactobacillary grade greater than 2 (LBG) (according to Donders classification);
* Vaginal dysbiosis based on microbial cell count.

Exclusion Criteria:

* Presence of sexually transmitted diseases due to Chlamydia, Neisseria gonorrhoeae or Trichomonas vaginalis as well as specific cervico-vaginitis or severe vulvovaginal symptoms related to acute candidiasis;
* Clinically evident herpes simplex infection;
* Human papillomavirus or human immunodeficiency virus infections;
* Use of antibiotics, antifungals, probiotics, or immunosuppressants within the past four weeks;
* Use of vaginal contraceptives and any other physiological or pathological condition that could potentially interfere with the results of the study (e.g. pregnancy or breastfeeding, chronic diseases, neoplastic diseases, diabetes, genital tract hemorrhages);
* Enrollment in other programs that involve the administration of products that may affect the composition of the vaginal microbiota.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women under reproductive age
Enrollment: 200 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Microbiota | Baseline; end of the treatment (10 days); wash-out (30 days)
  Change in the composition of the vaginal microbiota (significant reduction of pathogens responsible for vaginal dysbiosis and concomitant increase in lactobacilli)
Symptomatology | Baseline; end of the treatment (10 days); wash-out (30 days)
  Change of signs (leucorrhoea, vulvovaginal erythema/edema) and symptoms (vulvar discomfort, burning, itching) associated to vaginal dysbiosis. Clinical signs and symptoms will be evaluated through a severity score on a scale of 0 (absent or normal) to 3 (severe).
Sign | Baseline; end of the treatment (10 days); wash-out (30 days)
  Absence of inflammation according to Amsel's criteria and Nugent score between 0 and 3

SECONDARY OUTCOMES:
Well-being | Baseline and wash-out (30 days)
  Change in the quality of life, based on the Short Form-36 (SF-36) questionnaire. Values ranging from 0 to 100 indicate worst and better outcomes, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Palumbo, Prof, Study Director — University of Catania
Locations (1):
- University of Catania, Catania, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pino A, Vaccalluzzo A, Cianci S, Palumbo M, Caruso G, Caggia C, Randazzo CL. Oral Administration of the Probiotic Lacticaseibacillus rhamnosus CA15 in a Large Cohort of Women with Bacterial Vaginosis and Mixed Vaginitis: Clinical Evidence from a Randomized, Double-Blind, Placebo-Controlled Study. Microorganisms. 2025 Nov 21;13(12):2651. doi: 10.3390/microorganisms13122651. PMID 41471856